CLINICAL TRIAL: NCT06041633
Title: Preliminary Assessment of the Psycho-emotional State of Patients With TMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Malgorzata Pihut, Prof. Małgorzata Pihut, Jagiellonian University
Other Study IDs: 1072.6120.312.2021-15.12.2
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: C05.500.607.221.897; C05.550.905

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical: One hundred and thirty patients diagnosed with TMD constituted the study group (group I)
  Interventions: Diagnostic Test: Clinical
- Control: One hundred and thirty patients were excluded from having TMD based on the RDC/ TMD questionnaire, and these patients constituted the control group (group II).
  Interventions: Diagnostic Test: Clinical

INTERVENTIONS:
Diagnostic Test: Clinical — Questionnaire

SUMMARY:
TMD (temporomandibular disorders) is the name for a collective syndrome of disorders that includes abnormal function of the muscles of mastication, the temporomandibular joints and surrounding structures. It is one of the most significant causes of orofacial pain, along with dental pain. In TMD syndrome, the cause of pain is often due to overloading of the masticatory muscles rather than primary changes in the joints themselves.

Nowadays, doctors who treat patients with TMD have no doubt that one of the very important etiological factors of this condition is psycho-emotional disorders (excessive nervous excitability, anxiety, depression), which has been confirmed by numerous authors of studies on this subject [4-11].

The etiology of TMD is complex and multifactorial. Numerous factors may also contribute to the development of the disorder. An important factor affecting the state of masticatory function is an increase in stress levels (psycho-emotional tension). Structures such as the hypothalamus, reticular formation and limbic system have a decisive influence on the emotional state of each patient The activity of the limbic system, which governs the emotions of adults, and the additional connections of the gamma loops to the masticatory muscles, determine that increased emotional tension translates into a significant increase in the "contractile" activity of the masticatory muscles.

TMD and functional disorder of the masticatory muscles are the most common complaint of the patients, seeking treatment in dental office. The two main symptoms of TMD problems are pain and dysfunction. Myalgia -the most common cause is an increased level of muscle use. It is related to vasocontraction of relevant arteries and accumulation of metabolic waste product in the muscles. Activities such as daytime clenching of the teeth and bruxism, habits of chewing gum, biting lips, finger nails or cheeks are factors that cause significant strain on the masticatory muscles and temporomandibular joints.

ELIGIBILITY:
Inclusion Criteria:

(i) good general health, with no craniofacial trauma in the last 5 years and without severe mental conditions (ii) the presence of TMD symptoms (pain in the masticatory muscles, limitation of mouth opening range, clicking or popping in the temporomandibular joints. For control group there was absences of these symptoms.

(iii) consent of the patient to participate in the research project

The exclusion criteria for the study were:

-

Exclusion Criteria:

(i). willingness to resign out of the study.

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Population of Patients of University Clinic
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Questionanire | 2021-2023
  The questionnaire survey includes a total of 30 questions, regarding the emotional state of the of the respondents over the past 4 weeks such as lowered mood, states of emotional irritability, feelings of sadness, lack of desire for daily activities, lack of concentration, or desire for self-isolation and critical thoughts toward one's own person person, or nervousness, fearfulness. Responses in each question included: * no, * a few times in the past 4 weeks, *a few times during the week, and *continuously/continually. The scores for each question were: 0 points for most favorable response and 4 points for the most unfavorable patient response. The result of the questionnaire was divided into four sections; A, B, C,D.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersytecka Klinika Stomatologiczna, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pihut ME, Kostrzewa-Janicka J, Orczykowska M, Bieganska-Banas J, Gibas-Stanek M, Gala A. Initial assessment of the psycho-emotional state of patients with temporomandibular disorders: A pilot study. Dent Med Probl. 2024 Jan-Feb;61(1):153-159. doi: 10.17219/dmp/178325. PMID 38441313